CLINICAL TRIAL: NCT04017390
Title: The Effect of Theraworx Foam on the Cross-sectional Area of the Median Nerve in Patients With Carpal Tunnel Syndrome
Brief Title: The Effect of Theraworx Foam in Carpal Tunnel Syndrome
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of Funding from Sponsor
Sponsor: John Fowler (Other)
Collaborators: Avadim Technologies, Inc. (Industry)
Responsible Party: Sponsor-Investigator, John Fowler, Assistant Professor Department of Orthopaedic Surgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY19040180
Record Dates: First submitted 2019-07-04; First posted 2019-07-12 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Hand Pain/Numbness
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: Randomization will be to one of four groups: 1.) Theraworx foam alone; 2.) Theraworx foam plus night time splint; 3.) Placebo foam alone; 4.) Placebo foam plus night time splint.
  Theraworx Foam is an FDA registered (NDC 61594-001-02) topical agent (active ingredient: magnesium sulfate superficia 6 x 0.05% HPUS) for muscle cramp and spasm relief.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1: Theraworx Foam alone (Experimental): Theraworx foam only
  Interventions: Drug: Theraworx Foam
- Arm 2: Theraworx Foam and night splint (Active Comparator): Theraworx foam with a night time splint
  Interventions: Other: Theraworx Foam and night splint
- Arm 3: Placebo foam alone (Placebo Comparator): Placebo foam alone
  Interventions: Drug: Placebo Foam
- Arm 4: Placebo foam and night splint (Other): Placebo foam with a night time splint
  Interventions: Other: Placebo Foam and night time splint

INTERVENTIONS:
Drug: Theraworx Foam — Apply Theraworx Foam alone
  Arms: Arm 1: Theraworx Foam alone
Drug: Placebo Foam — Apply placebo foam alone
  Arms: Arm 3: Placebo foam alone
Other: Theraworx Foam and night splint — Apply Theraworx Foam and night time splint
  Arms: Arm 2: Theraworx Foam and night splint
Other: Placebo Foam and night time splint — Apply placebo foam and night time splint
  Arms: Arm 4: Placebo foam and night splint

SUMMARY:
Participation will be for approximately 21 days (3 study visits,1 week apart with allowance for scheduling conflicts). A topical (or placebo) foam alone or with a splint will be used. Demographic and symptom information will be obtained. At each visit 3 questionnaires (BCT, CTS-6, and DASH) will be completed and an ultrasound of the wrist (median nerve) will be done to document any change in symptoms and/or in the size of the nerve. Random assignment will be to one of 4 groups: foam or placebo with or without a night splint. We will provide instruction on how to apply the foam, whether or not and how to wear the splint, and return visits.

DETAILED DESCRIPTION:
The PI will identify potential participants from his clinical practice. Evaluation of symptoms will be by exam, questionnaires, and ultrasound of the median nerve. These will document baseline/change in the size of the median nerve and improvement in function/symptoms. The questionnaires are 1.) Boston Carpal Tunnel (BCT). 2.) Carpal Tunnel-6 (CTS-6); and 3.) Disabilities of the Arm, Shoulder and Hand (DASH). These will be used to document a baseline and change (if any) in nerve size and hand symptoms, over a 2 week time frame, that are common in carpal tunnel syndrome (including numbness, pain, tingling, and/or decreased function).

1. The Boston Carpal Tunnel is a 19 question tool that assesses function (8 items) and symptom severity (11 items). Score range is from 0 to 95 with a high number indicating more severe/worsening symptoms and lower number less severe/improving symptoms.
2. The CTS-6 is a six item tool that combines reported symptoms with a physical exam of the hand. Scores range from 0 to 26 with a higher score reflecting increased severity.
3. The DASH is a 30 item tool with each scored 1 to 5. Scores can range from 0 to 150 and the higher the score the worse the symptoms/disability.

Treatment groups are as follows:1.) Theraworx foam alone; 2.) Theraworx foam with night time splint; 3.) Placebo foam alone; 4.) Placebo foam with night time splint. The active ingredient in Theraworx foam is magnesium sulfate and will not be in the placebo foam. Instructions on how to apply the foam, whether or not and how to wear the splint, and return visits will be provided. If in a group that requires night time splinting, the subject must wear the splint only at night and for a minimum of 8 hours.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Carpal Tunnel Syndrome
* Age 18 years or older
* Interest in non-surgical treatment of carpal tunnel syndrome

Exclusion Criteria:

* Prior carpal tunnel release
* Non-English speaking
* Skin lesions/rashes on hand being treated
* Current use of topical anti-inflammatory medication
* Other diagnoses that would impact results (determined by PI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-01-03 (Actual); Study Completion 2022-01-03 (Actual)

PRIMARY OUTCOMES:
Improvement (decrease) in size of median nerve at the wrist | 2 weeks
  Decrease in cross sectional area of median nerve as determined by ultrasound exam

SECONDARY OUTCOMES:
Improvement (decrease) in Boston Carpal Tunnel Questionnaire (BCTQ) | 2 weeks
  Improvement in PRO as indicated by a decreased score on questionnaire indicating improved in function and decreased symptoms
Improvement (decrease) in Carpal Tunnel 6 (CTS-6) score | 2 weeks
  Improvement in patient reported outcome (PRO) as determined by a lower CTS-6 score number than at baseline. Score ranges from 26 (worst) to 0 (best)
Improvement (decrease) in Disabilities of Arm, Shoulder, Hand (DASH) score | 2 weeks
  Improvement in patient reported outcome (PRO) as determined by decreased DASH score from baseline. Score ranges from 150 (worst) to 30 (best)

CONTACTS AND LOCATIONS:
Overall Officials: John Fowler, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Kaufmann Building, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The ultrasound measurements and PRO questionnaire scores will be shared with the sponsor Avadim Technologies at a minimum of approximately 60 day intervals throughout the study (1 year) and at the discretion of the PI. In addition, final data will be provided within 12 months of completion of last participant
Supporting Information: Study Protocol, CSR
Time Frame: Updated at intervals of approximately 60 days (minimum) and as needed as determined by PI. Final data will be available approximately 12 months after completion of last participant and will be available for 9 to 12 months.